CLINICAL TRIAL: NCT05218395
Title: Association Between Persistent Organic Pollutants and Type 2 Diabetes /Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: YXLL-KY-2021(064)
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes; Thyroid Cancer; Organic Pollutant
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Persistent organic pollutants (POPs) are a class of organic pollutants in the environment characterized by persistent, bioaccumulation, long-range transport and biological toxicity. Due to its widespread distribution in the environment and Lipophilicity, POPs can bioaccumulate along the food chain and eventually accumulate in the human body. There are many types of POPs, including dioxins, polychlorinated biphenyls (PCBs) , polybrominated diphenyl ethers (PBDEs) and organochlorine pesticides (OCPs) . POPs is ubiquitous and Lipophilic in the environment, so the potential harm of POPs to human body has aroused wide concern. A growing number of studies have found that exposure to POPs may be associated with an increased risk of endocrine disease, particularly type 2 diabetes and thyroid cancer.

The aim of this study was to assess the effect of Persistent organic pollutant exposure on the development ofType 2 diabetes and thyroid cancer by analyzing serum Persistent organic pollutant concentrations in controls, and patients with Type 2 diabetes and thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

Group of Type 2 diabetes patients:

1. age 18 ~ 75 years old;
2. type 2 diabetes patients diagnosed in the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province) , HBA1C ≥7.0% and <10.5% ;
3. patients signed informed consent.

Group of Thyroid Cancer patients:

1. age 18 ~ 75 years old;
2. thyroid cancer patients diagnosed in the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province) ;
3. patients who signed the informed consent form.

Control Group:

1. age 18 ~ 75 years old;
2. healthy population recruited from the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province) ;
3. living in the monitoring area for more than 6 months within 12 months;
4. normal thyroid function and no history of thyroid cancer were needed in the control group;
5. Fasting Blood Glucose level of 0.7 mmol/l was needed in the Control Group of Type 2 diabetes Mellitus Without History of diabetes;
6. patients with informed consent.

Exclusion Criteria:

* Group of Type 2 diabetes:

  (1) pregnant, lactating women, patients with acute cardiac cerebrovascular disease; (2) patients with severe liver and Renal Impairment (related laboratory tests more than 2 times the normal) ; (3) patients with Type 1 diabetes; (4) participants in other clinical trials within 3 months; (5) patients with malignant tumors. (6) has the disease and so on serious anemia, is not suitable to carry on the patient which the blood draws the test.

Group of Thyroid Cancer:

1. patients with serious heart, liver and Kidney Diseases (related laboratory tests more than 2 times normal) ;
2. patients with other malignant tumors.

Control Group:

1. patients with serious heart, liver or kidney disease;
2. patients with iodine or Thyroid hormone;
3. patients with confirmed malignant tumor;
4. pregnant women or those who have recently taken contraception or estrogen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population：18 ~ 75 years old patients of type 2 diabetes，Thyroid Cancer and control。
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the risk of Persistent organic pollutant exposure to type 2 diabetes | 2021．11 Ethics Committee Approval 2021.12-2024.12 controls/patients recruitment, samples test 2025.1-2024.12 data analysis
  to explore the effect of Persistent organic pollutant on the risk of type 2diabetes

SECONDARY OUTCOMES:
To assess the risk of Persistent organic pollutant exposure to thyroid cancer | 2021．11 Ethics Committee Approval 2021.12-2024.12 controls/patients recruitment, samples test 2025.1-2024.12 data analysis
  to explore the effect of Persistent organic pollutant on the risk of thyroid cancer

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Guan, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Xiaoling Guan, Jinan, Shandong, China